CLINICAL TRIAL: NCT02084368
Title: Application of Combined Lumbar Plexus and Sciatic Nerve Block in Unilateral Knee Replacement
Brief Title: Application of Combined Lumbar Plexus and Sciatic Nerve Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, bo xu, associate chief physician, Guangzhou General Hospital of Guangzhou Military Command
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nerve Block
Record Dates: First submitted 2014-03-06; First posted 2014-03-12 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Anesthesia
Keywords: combined lumbar plexus and sciatic nerve block，; combined spinal and epidural anesthesia
MeSH Terms: interventions — Nerve Block; Anesthesia, Epidural; Ropivacaine; Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nerve block (Experimental): Patients in this group were assigned to receive lumbar plexus block and sciatic nerve block guided by PNS.
  Interventions: Procedure: Nerve block; Drug: Ropivacaine
- combined spinal and epidural anesthesia (Placebo Comparator): Combined spinal and epidural anesthesia were performed in patients of this group.
  Interventions: Procedure: Combined spinal and epidural anesthesia; Drug: Bupivacaine

INTERVENTIONS:
Procedure: Nerve block — Patients in this group were assigned to receive lumbar plexus block and sciatic nerve block both using 0.33% ropivacaine 30ml guided by PNS
  Arms: Nerve block
Procedure: Combined spinal and epidural anesthesia — Combined spinal and epidural anesthesia were performed in patients of this group with 0.5% hyperbaric bupivacaine 8~10mg at L2-3 or L3-4.
  Arms: combined spinal and epidural anesthesia
Drug: Ropivacaine — Patients will be assigned to receive lumbar plexus block and sciatic nerve block both using 0.33% ropivacain 30ml guided by PNS.
  Other Names: 0.33%Ropivacaine
  Arms: Nerve block
Drug: Bupivacaine — Combined spinal and epidural anesthesia will be performed in patients with 0.5% hyperbaric bupivacaine 8~10mg.
  Other Names: 0.5%Bupivacaine
  Arms: combined spinal and epidural anesthesia

SUMMARY:
The research is to study the effectiveness and safety of combined lumbar plexus and sciatic nerve block by the guide of peripheral nerve stimulator (PNS) in unilateral knee replacement.There have be some papers which supported that combined lumbar plexus and sciatic nerve block may be more suitable for the old men.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of American Association of anesthetists（ASA）Grade 1、2 or 3
2. Aged between 18 and 85 years
3. Undergoing elective total knee replacement.

Exclusion Criteria:

1. Mental illness can not match
2. Nerve block, epidural anesthesia contraindicated
3. People who have Slow-type arrhythmias
4. History of chronic headaches and long-term use of analgesic drugs
5. People who were postoperative consciousness, language or hearing impaired

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Maintenance time of sensory and motor nerve block | up to 24h after operation
  from the end of injection of local anesthetic drug up to 24h after operation

SECONDARY OUTCOMES:
The change of hemodynamics | 0, 5, 10, 20, 30, 60 min after injection
  the changes of SBP and DBP at 0, 5, 10, 20, 30, 60 min after injection

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Military Region General Hospital, Department of Anesthesiology, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Farny J, Girard M, Drolet P. Posterior approach to the lumbar plexus combined with a sciatic nerve block using lidocaine. Can J Anaesth. 1994 Jun;41(6):486-91. doi: 10.1007/BF03011542. PMID 8069988
- [Result] de Leeuw MA, Slagt C, Hoeksema M, Zuurmond WW, Perez RS. Hemodynamic changes during a combined psoas compartment-sciatic nerve block for elective orthopedic surgery. Anesth Analg. 2011 Mar;112(3):719-24. doi: 10.1213/ANE.0b013e318206bc30. Epub 2010 Dec 14. PMID 21156977